CLINICAL TRIAL: NCT06797804
Title: Effectiveness of Information Technology-Assisted Horticultural Therapy Program on Heart Rate Variability, Stress, Depression and Happiness Among Older Adults Resident in Long-Term Care Facilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph. D, RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKH-IRB-20240809R
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Heart Rate Variability; Stress; Depression; Happiness
Keywords: Horticultural Therapy; Older adults; Information and communication technology; Mental health
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Horticultural Therapy

STUDY DESIGN:
Intervention Model Description: cluster-randomized controlled trial，cRCT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Information Technology-Assisted Horticultural Therapy Program (Experimental): The intervention involves technology-assisted horticultural therapy sessions conducted once a week, lasting 120 minutes per session, over a total period of 8 weeks.
  Interventions: Other: Information Technology-Assisted Horticultural Therapy Program
- Routine Care (No Intervention): No intervention will be applied to the routine care group.

INTERVENTIONS:
Other: Information Technology-Assisted Horticultural Therapy Program — The intervention involves technology-assisted horticultural therapy sessions conducted once a week, lasting 120 minutes per session, over a total period of 8 weeks
  Other Names: Horticultural Therapy; Horticultural activity; horticultural intervention
  Arms: Information Technology-Assisted Horticultural Therapy Program

SUMMARY:
This study aims to address existing research gaps by investigating the effects of technology-assisted horticultural therapy on stress, depression, and happiness among older adults residing in long-term care facilities. By examining the modulation of the autonomic nervous system, the findings will provide a foundation for developing comprehensive health promotion programs that integrate traditional therapeutic practices with modern technology to enhance the well-being of the aging population.

DETAILED DESCRIPTION:
The mental health needs of older adults are a growing concern, and as technology advances, integrating health information with technology can improve healthcare quality and dissemination efficiency. Integrating health information with technology holds promise for enhancing healthcare quality and dissemination efficiency in practical applications, thereby equipping more individuals with accurate health maintenance knowledge. Particularly notable is the increasing trend in internet usage among modern seniors, which contributes to achieving United Nations Sustainable Development Goals. Horticultural therapy has been widely acknowledged for its positive impact on human well-being in various settings. However, its integration with information technology remains relatively unexplored. Additionally, studies on its effectiveness in relieving stress have demonstrated inconsistent effects on heart rate variability. Therefore, this study aims to examine how technology-assisted horticultural therapy influences stress, depression, and happiness among older adult residents in long-term care facilities, with a specific focus on regulating the autonomic nervous system. The study will employ both subjective questionnaire surveys and objective measurements of heart rate. This study proposes a cluster randomized controlled trial. Using G-Power 3.1, a minimum sample size of 76 participants is calculated, accounting for an estimated 20% attrition rate. To ensure equitable distribution between intervention and control groups, each group will consist of at least 38 participants. The intervention involves technology-assisted horticultural therapy sessions conducted once a week, lasting 120 minutes per session, over a total period of 8 weeks. The research will employ several tools: (1) a basic demographic questionnaire, (2) the Mini-Mental State Examination (MMSE), (3) the 'Taiwan Scientific' Noninvasive Blood Pressure Meter (TS 0411), (4) the Perceived Stress Scale (PSS), (5) the Geriatric Depression Scale (GDS-15), and (6) the 5-item World Health Organization Well-Being Index (WHO-5). Data collection will span pre-, mid-, and post-intervention periods over 8 weeks for both experimental and control groups. The Efficacy of Horticultural Therapy Evaluation Form (EHTE) will also be used to conduct pre-test and post-test evaluations on the experimental group. Data will be analyzed using SPSS 27.0. Descriptive statistics will be applied to the demographic questionnaire data, while generalized estimating equations (GEE) will analyze pre-, mid-, and post-test questionnaire responses and objective measurements. Empirical evidence from this study will elucidate the impact of technology-assisted horticultural therapy on heart rate variability, stress, depression, and happiness among older adult residents in long-term care facilities. These findings will serve as a basis for developing health pro-motion programs aimed at enhancing the physical and mental well-being of aging populations.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this study
2. Elderly persons aged 65 and above living in long-term care facilities
3. Live in long-term care facilities for at least three months
4. No gender restrictions
5. Be aware, able to communicate in Mandarin and Taiwanese, and be able to express opinions
6. The upper limbs can move freely and there is no disease that causes tremors in the hands (such as Parkinson's disease, hepatic encephalopathy, etc.)

Exclusion Criteria:

1. Has participated in gardening-related activities within one month of receiving the case
2. Those diagnosed with terminal illness or whose health condition is rapidly deteriorating
3. Those suffering from Parkinson's disease, serious heart disease, dementia, mental illness (e.g. schizophrenia, bipolar disorder, etc.)
4. Mini-Mental State Examination (MMSE) with cognitive impairment (MMSE scores below 16 points for individuals with no formal education, below 21 points for those with elementary education, and below 24 points for those with junior high school education or higher.)
5. Those who are unable to participate in the event due to severe speech, vision or hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability, HRV | Baseline, pre-intervention (T0)
  The most frequently used method for Autonomic Nervous System (ANS) test. Heart rate variability (HRV) represents total activity index of ANS; The higher the HRV, the better the ANS control.
Perceived Stress Scale, PSS | Baseline, pre-intervention (T0)
  The total score serves as an overall indicator of stress levels. It demonstrates good internal reliability, with a Cronbach's alpha coefficient of 0.85. The scale comprises 14 items, the total score ranges from 0 to 56, with higher scores indicating greater perceived stress.
Geriatric Depression Scale, GDS-15 | Baseline, pre-intervention (T0)
  The Geriatric Depression Scale (GDS) is a widely used screening tool designed to identify depression in older adults. The GDS-15 has been translated and adapted for use in various cultural contexts, including Chinese-speaking populations. The scale demonstrated good reliability (Cronbach's α = .94). The total score ranging from 0 to 15. The higher scores indicate greater severity of depressive symptoms.
The 5-item World Health Organization Well-Being Index, WHO-5 | Baseline, pre-intervention (T0)
  The WHO-5 Well-Being Index is a brief, universally applicable global scale for measuring subjective well-being. The scale consists of five items, each scored from 0 to 5. The raw score ranges from 0 to 25, with higher scores indicating greater well-being. The raw score is often multiplied by 4 to convert it to a percentage scale ranging from 0 to 100.
The efficacy of horticultural therapy evaluation form; EHTE | Baseline, pre-intervention (T0)
  The scale used to measure the well-being gained from horticultural therapy defines well-being as a state where an individual can demonstrate their abilities, cope with daily stress, be effective and productive at work, and contribute to society. The Cronbach's α value was 0.724, indicating good reliability. The total score ranging from 7 to 35. The higher the score and the larger the difference between pre- and post-tests, the greater the well-being gained by participants in the horticultural therapy.
Heart Rate Variability, HRV | 4 weeks after intervention (T1)
  The most frequently used method for Autonomic Nervous System (ANS) test. Heart rate variability (HRV) represents total activity index of ANS; The higher the HRV, the better the ANS control.
Perceived Stress Scale, PSS | 4 weeks after intervention (T1)
  The total score serves as an overall indicator of stress levels. It demonstrates good internal reliability, with a Cronbach's alpha coefficient of 0.85. The scale comprises 14 items, the total score ranges from 0 to 56, with higher scores indicating greater perceived stress.
Geriatric Depression Scale, GDS-15 | 4 weeks after intervention (T1)
  The Geriatric Depression Scale (GDS) is a widely used screening tool designed to identify depression in older adults. The GDS-15 has been translated and adapted for use in various cultural contexts, including Chinese-speaking populations. The scale demonstrated good reliability (Cronbach's α = .94). The total score ranging from 0 to 15. The higher scores indicate greater severity of depressive symptoms.
The 5-item World Health Organization Well-Being Index, WHO-5 | 4 weeks after intervention (T1)
  The WHO-5 Well-Being Index is a brief, universally applicable global scale for measuring subjective well-being. The scale consists of five items, each scored from 0 to 5. The raw score ranges from 0 to 25, with higher scores indicating greater well-being. The raw score is often multiplied by 4 to convert it to a percentage scale ranging from 0 to 100.
Heart Rate Variability, HRV | 8 weeks after intervention (T2)
  The most frequently used method for Autonomic Nervous System (ANS) test. Heart rate variability (HRV) represents total activity index of ANS; The higher the HRV, the better the ANS control.
Perceived Stress Scale, PSS | 8 weeks after intervention (T2)
  The total score serves as an overall indicator of stress levels. It demonstrates good internal reliability, with a Cronbach's alpha coefficient of 0.85. The scale comprises 14 items, the total score ranges from 0 to 56, with higher scores indicating greater perceived stress.
Geriatric Depression Scale, GDS-15 | 8 weeks after intervention (T2)
  The Geriatric Depression Scale (GDS) is a widely used screening tool designed to identify depression in older adults. The GDS-15 has been translated and adapted for use in various cultural contexts, including Chinese-speaking populations. The scale demonstrated good reliability (Cronbach's α = .94). The total score ranging from 0 to 15. The higher scores indicate greater severity of depressive symptoms.
The 5-item World Health Organization Well-Being Index, WHO-5 | 8 weeks after intervention (T2)
  The WHO-5 Well-Being Index is a brief, universally applicable global scale for measuring subjective well-being. The scale consists of five items, each scored from 0 to 5. The raw score ranges from 0 to 25, with higher scores indicating greater well-being. The raw score is often multiplied by 4 to convert it to a percentage scale ranging from 0 to 100.
The efficacy of horticultural therapy evaluation form; EHTE | 8 weeks after intervention (T2)
  The scale used to measure the well-being gained from horticultural therapy defines well-being as a state where an individual can demonstrate their abilities, cope with daily stress, be effective and productive at work, and contribute to society. The Cronbach's α value was 0.724, indicating good reliability. The total score ranging from 7 to 35. The higher the score and the larger the difference between pre- and post-tests, the greater the well-being gained by participants in the horticultural therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marioni RE, Chatfield M, Brayne C, Matthews FE; Medical Research Council Cognitive Function and Ageing Study Group. The reliability of assigning individuals to cognitive states using the Mini Mental-State Examination: a population-based prospective cohort study. BMC Med Res Methodol. 2011 Sep 6;11:127. doi: 10.1186/1471-2288-11-127. PMID 21896187
- [Background] Ng KST, Sia A, Ng MKW, Tan CTY, Chan HY, Tan CH, Rawtaer I, Feng L, Mahendran R, Larbi A, Kua EH, Ho RCM. Effects of Horticultural Therapy on Asian Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Aug 9;15(8):1705. doi: 10.3390/ijerph15081705. PMID 30096932
- [Background] Park, S., Lee, A., Son, K., Lee, W., & Kim, D. (2016). Gardening Intervention for Physical and Psychological Health Benefits in Elderly Women at Community Centers. HortTechnology hortte, 26(4), 474-483. https://doi.org/10.21273/HORTTECH.26.4.474
- [Background] Sheikh, J.I. and Yesavage, J.A. (1986) Geriatric Depression Scale (GDS): Recent Evidence and Development of a Shorter Version. Clinical Gerontologist: The Journal of Aging and Mental Health, 5, 165-173. https://doi.org/10.1300/J018v05n01_09
- [Background] Todd RM, Miskovic V, Chikazoe J, Anderson AK. Emotional Objectivity: Neural Representations of Emotions and Their Interaction with Cognition. Annu Rev Psychol. 2020 Jan 4;71:25-48. doi: 10.1146/annurev-psych-010419-051044. Epub 2019 Oct 14. PMID 31610131
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Tsai YI, Beh J, Ganderton C, Pranata A. Digital interventions for healthy ageing and cognitive health in older adults: a systematic review of mixed method studies and meta-analysis. BMC Geriatr. 2024 Mar 4;24(1):217. doi: 10.1186/s12877-023-04617-3. PMID 38438870
- [Background] Tu PC, Cheng WC, Hou PC, Chang YS. Effects of Types of Horticultural Activity on the Physical and Mental State of Elderly Individuals. Int J Environ Res Public Health. 2020 Jul 20;17(14):5225. doi: 10.3390/ijerph17145225. PMID 32698351
- [Background] Vassanyi I, Szakonyi B, Loi D, Mantur-Vierendeel A, Quintas J, Solinas A, Blazica B, Raffo L, Guicciardi M, Manca A, Gaal B, Rarosi F. Impact of information technology supported serious leisure gardening on the wellbeing of older adults: The Turntable project. Geriatr Nurs. 2024 Jan-Feb;55:339-345. doi: 10.1016/j.gerinurse.2023.12.014. Epub 2023 Dec 29. PMID 38159476
- [Background] Yeo NL, Elliott LR, Bethel A, White MP, Dean SG, Garside R. Indoor Nature Interventions for Health and Wellbeing of Older Adults in Residential Settings: A Systematic Review. Gerontologist. 2020 Apr 2;60(3):e184-e199. doi: 10.1093/geront/gnz019. PMID 30884495
- [Background] Luppa M, Luck T, Weyerer S, Konig HH, Brahler E, Riedel-Heller SG. Prediction of institutionalization in the elderly. A systematic review. Age Ageing. 2010 Jan;39(1):31-8. doi: 10.1093/ageing/afp202. Epub 2009 Nov 23. PMID 19934075
- [Background] Luk KY, Lai KY, Li CC, Cheung WH, Lam SM, Li HY, Ng KP, Shiu WH, So CY, Wan SF. The effect of horticultural activities on agitation in nursing home residents with dementia. Int J Geriatr Psychiatry. 2011 Apr;26(4):435-6. doi: 10.1002/gps.2493. No abstract available. PMID 21412848
- [Background] Lin TY, Huang CM, Hsu HP, Liao JY, Cheng VY, Wang SW, Guo JL. Effects of a Combination of Three-Dimensional Virtual Reality and Hands-on Horticultural Therapy on Institutionalized Older Adults' Physical and Mental Health: Quasi-Experimental Design. J Med Internet Res. 2020 Nov 2;22(11):e19002. doi: 10.2196/19002. PMID 33135666
- [Background] Lai, P. Y., Chen, C.H. (2017). Design an Interactive Game App of Horticultural Therapy for Older Adults. In: Hale, K., Stanney, K. (eds) Advances in Neuroergonomics and Cognitive Engineering. Advances in Intelligent Systems and Computing, 488. Springer, Cham. https://doi.org/10.1007/978-3-319-41691-5_35
- [Background] Lai CKY, Kwan RYC, Lo SKL, Fung CYY, Lau JKH, Tse MMY. Effects of Horticulture on Frail and Prefrail Nursing Home Residents: A Randomized Controlled Trial. J Am Med Dir Assoc. 2018 Aug;19(8):696-702. doi: 10.1016/j.jamda.2018.04.002. Epub 2018 May 24. PMID 29804892
- [Background] Kim Y, Hong S, Choi M. Effects of Serious Games on Depression in Older Adults: Systematic Review and Meta-analysis of Randomized Controlled Trials. J Med Internet Res. 2022 Sep 6;24(9):e37753. doi: 10.2196/37753. PMID 36066964
- [Background] Hung YC, Chen YH, Lee MC, Yeh CJ. Effect of Spousal Loss on Depression in Older Adults: Impacts of Time Passing, Living Arrangement, and Spouse's Health Status before Death. Int J Environ Res Public Health. 2021 Dec 10;18(24):13032. doi: 10.3390/ijerph182413032. PMID 34948641
- [Background] Hou CJ, Chen YT, Capilayan M, Lin YS, Huang MW, Huang JJ. Analysis of Heart Rate Variability in Response to Serious Games in Elderly People. Sensors (Basel). 2021 Sep 30;21(19):6549. doi: 10.3390/s21196549. PMID 34640863
- [Background] Han AR, Park SA, Ahn BE. Reduced stress and improved physical functional ability in elderly with mental health problems following a horticultural therapy program. Complement Ther Med. 2018 Jun;38:19-23. doi: 10.1016/j.ctim.2018.03.011. Epub 2018 Mar 28. PMID 29857876
- [Background] Guimaraes LA, Brito TA, Pithon KR, Jesus CS, Souto CS, Souza SJN, Santos TSD. Depressive symptoms and associated factors in elderly long-term care residents. Cien Saude Colet. 2019 Sep 9;24(9):3275-3282. doi: 10.1590/1413-81232018249.30942017. English, Portuguese. PMID 31508748
- [Background] Grolli RE, Mingoti MED, Bertollo AG, Luzardo AR, Quevedo J, Reus GZ, Ignacio ZM. Impact of COVID-19 in the Mental Health in Elderly: Psychological and Biological Updates. Mol Neurobiol. 2021 May;58(5):1905-1916. doi: 10.1007/s12035-020-02249-x. Epub 2021 Jan 6. PMID 33404981
- [Background] Gramaglia C, Gattoni E, Marangon D, Concina D, Grossini E, Rinaldi C, Panella M, Zeppegno P. Non-pharmacological Approaches to Depressed Elderly With No or Mild Cognitive Impairment in Long-Term Care Facilities. A Systematic Review of the Literature. Front Public Health. 2021 Jul 16;9:685860. doi: 10.3389/fpubh.2021.685860. eCollection 2021. PMID 34336772
- [Background] Giunti G, Baum A, Giunta D, Plazzotta F, Benitez S, Gomez A, Luna D, Bernaldo de Quiros FG. Serious Games: A Concise Overview on What They Are and Their Potential Applications to Healthcare. Stud Health Technol Inform. 2015;216:386-90. PMID 26262077
- [Background] Fan CC, Choy CS, Huang CM, Chih PS, Lee CC, Lin FH, Guo JL. The effects of a combination of 3D virtual reality and hands-on horticultural activities on mastery, achievement motives, self-esteem, isolation and depression: a quasi-experimental study. BMC Geriatr. 2022 Sep 12;22(1):744. doi: 10.1186/s12877-022-03431-7. PMID 36096746
- [Background] Ernst H, Scherpf M, Pannasch S, Helmert JR, Malberg H, Schmidt M. Assessment of the human response to acute mental stress-An overview and a multimodal study. PLoS One. 2023 Nov 9;18(11):e0294069. doi: 10.1371/journal.pone.0294069. eCollection 2023. PMID 37943894
- [Background] Chou HC, Cheng SF, Jennifer Yeh SC, Tang PL. Effectiveness of a multicomponent activity and horticultural intervention for the hospitalized older adults: A randomized controlled trial: Effectiveness of Intervention for the Hospitalized Older Adults. Geriatr Nurs. 2024 Jan-Feb;55:112-118. doi: 10.1016/j.gerinurse.2023.10.024. Epub 2023 Nov 17. PMID 37979470
- [Background] Bautista TG, Roman G, Khan M, Lee M, Sahbaz S, Duthely LM, Knippenberg A, Macias-Burgos MA, Davidson A, Scaramutti C, Gabrilove J, Pusek S, Mehta D, Bredella MA. What is well-being? A scoping review of the conceptual and operational definitions of occupational well-being. J Clin Transl Sci. 2023 Oct 16;7(1):e227. doi: 10.1017/cts.2023.648. eCollection 2023. PMID 38028344
- [Background] Lu S, Liu J, Xu M, Xu F. Horticultural therapy for stress reduction: A systematic review and meta-analysis. Front Psychol. 2023 Jul 26;14:1086121. doi: 10.3389/fpsyg.2023.1086121. eCollection 2023. PMID 37564307